CLINICAL TRIAL: NCT04776135
Title: A Phase I, Randomized, Open-Label, Crossover-Design, Single-Dose Study to Investigate the Safety, Tolerability and Comparative Bioavailability of Oral Edaravone Administered Orally and Via a Nasogastric Tube (NGT) in Healthy Adult Subjects
Brief Title: Comparative Bioavailability Study of Oral Edaravone Administered Orally and Via a Nasogastric Tube
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MT-1186-Z-101; jRCT2031200361 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — Edaravone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MT-1186 orally (Experimental): Subjects receive the edaravone oral suspension orally.
  Interventions: Drug: MT-1186
- MT-1186 via a nasogastric tube (Experimental): Subjects receive the edaravone oral suspension via a nasogastric tube
  Interventions: Drug: MT-1186

INTERVENTIONS:
Drug: MT-1186 — Suspension
  Other Names: Edaravone

SUMMARY:
To investigate the comparative bioavailability of edaravone oral suspension administered orally and via a nasogastric tube in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria: Subjects who meet all of the following criteria and who have the capability of giving informed consent will be included in the study.

1. Healthy adult male or female volunteers
2. Japanese
3. Subjects aged between 20 and 45 years at the time of informed consent
4. Subjects who have thoroughly understood the contents of the study and voluntarily provided written informed consent to participate in the study

Exclusion Criteria: Subjects who meet any of the following criteria between screening and investigational product administration will be excluded from the study.

1. Subjects with a current or previous history of cardiac, hepatic, renal, gastrointestinal, respiratory, psychiatric/nervous, hematopoietic, or endocrine diseases, and those whom the investigator (or subinvestigator) deems unsuitable for the study
2. History of drug or food allergies
3. History of alcohol or drug abuse or dependence
4. Body mass index (BMI) of <18.0 or >30.0, or a body weight of <50 kg (BMI formula: body weight [kg]/height [m]2, rounded to one decimal place)
5. Positive test for any of the following at screening: Hepatitis B surface antigen, serological test for syphilis, hepatitis C virus antibody, or human immunodeficiency virus antigen/antibody, subject has a positive COVID-19 virus test on Day -1
6. Any clinically significant 12-lead ECG abnormality or QTcF interval ≥450 msec
7. Blood donation or sampling with a total volume of ≥400 mL within 12 weeks, ≥200 mL within 4 weeks, or ≥800 mL within one year before providing informed consent
8. Blood component donation or blood sampling within 2 weeks before providing informed consent, or blood donation and transfusion from informed consent to the start of investigational product administration
9. Subjects who have undergone any surgery known to affect the gastrointestinal absorption of drugs (except for appendectomy and herniotomy)
10. Female subjects of childbearing potential who do not agree to use an effective method of contraception from screening or 2 weeks before the start of investigational product administration, whichever comes earlier, to 14 days after the completion (or discontinuation) of investigational product administration. Male subjects who do not agree to use an effective method of contraception from the start of investigational product administration to 14 days after the completion (or discontinuation) of investigational product administration
11. Subjects who have previously received edaravone
12. Subjects who have participated in another clinical study and received an investigational product within 12 weeks before providing informed consent
13. Subjects who have used any drugs other than the single use of acetylsalicylic acid within 7 days before the initiation of investigational product administration
14. Use of alcohol or any products containing xanthin or caffeine within 24 hours before screening and visit on Day -1
15. Use of any nutritional supplement(s) within 7 days before the initiation of investigational product administration
16. Use of grapefruit, grapefruit juice, or any processed food(s) containing these substances within 24 hours before screening and visit on Day -1
17. Use of any tobacco or nicotine-containing product(s) within 24 hours before screening and visit on Day -1
18. Female subjects who have a positive pregnancy test at screening and on Day -1, are pregnant or breast feeding, or plan to get pregnant during the study
19. Subjects with a history of reconstructive nasal surgery, or any evidence of deformities or asymmetry of the nose, non-patent nares/obstructed nasal airway, or the presence of nasal ulcers or polyps that would prevent an adequate NGT insertion.
20. Subjects judged by the investigator (or subinvestigator) to be unsuitable for the study for any other reason

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Investigational site, Tokyo, Toshima-ku, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shimizu H, Nishimura Y, Shiide Y, Ueda M, Yokota S, Kato Y, Hirai M. Edaravone Administered Orally and Via Nasogastric Tube in Healthy Adults: A Comparative Bioavailability Phase 1 Study. Clin Pharmacol Drug Dev. 2023 Jan;12(1):77-84. doi: 10.1002/cpdd.1175. Epub 2022 Oct 12. PMID 36225132

RESULTS

PARTICIPANT FLOW:
Groups:
- MT-1186 Orally, Then MT-1186 Via a Nasogastric Tube (NGT): Period 1: a single dose of Edaravone oral suspension orally. Period 2: a single dose of Edaravone oral suspension via a NGT.
- MT-1186 Via NGT, Then MT-1186 Orally: Period 1: a single dose of Edaravone oral suspension via NGT. Period 2 : a single dose of Edaravone oral suspension orally.
Period: Period 1
Arm/Group | MT-1186 Orally, Then MT-1186 Via a Nasogastric Tube (NGT) | MT-1186 Via NGT, Then MT-1186 Orally
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Period 2
Arm/Group | MT-1186 Orally, Then MT-1186 Via a Nasogastric Tube (NGT) | MT-1186 Via NGT, Then MT-1186 Orally
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MT-1186 Orally, Then MT-1186 Via a Nasogastric Tube (NGT) | MT-1186 Via NGT, Then MT-1186 Orally | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 12 | 12 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 18 | 18 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Versus Time Curve (AUC) of Edaravone
Description: Area under the plasma concentration versus time curve from time zero up to the last quantifiable concentration time-point (AUC0-t) of edaravone, and Area under the plasma concentration versus time curve from time zero up to infinity with extrapolation of the terminal phase (AUC0-inf) of edaravone.
Time Frame: Plasma samples are collected: Day 1 and Day 4 at pre-dose, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, and 12 hours; Day 2 and Day 5 at 24 and 36 hours; Day 3 and Day 6 at 48 hours after administration.
Population: This study was designed as a 2-group, 2-period crossover study with the advance administration of edaravone orally group (Oral => NGT) with 18 subjects, and the advance administration of edaravone via NGT group (NGT => Oral) with 18 subjects to investigate the bioavailability between edaravone orally and via NGT.
Measure: Mean (Standard Deviation); unit: ng·h/mL
Groups:
- MT-1186 Via NGT: Subjects receive the edaravone oral suspension via NGT
Arm/Group | MT-1186 Orally | MT-1186 Via NGT
Number analyzed (Participants) | 36 | 36
ng·h/mL
  AUC0-t | 2612 (787) | 2592 (866)
  AUC0-inf | 2657 (801) | 2617 (870)
Statistical Analysis 1: Comparison: MT-1186 Orally vs MT-1186 Via NGT; For AUC0-t, MT-1186 orally Versus MT-1186 via NGT; Test type: Other — AUC0-t was log-transformed and analyzed by analysis of variance using administration groups, the administration route, study periods, and subjects as factors. Estimates of the mean values on the log scale, the mean difference between administration routes on the log scale, and 90% CIs for the difference were back transformed to present mean ratios and their 90% CIs for administration via NGT to oral administration; ANOVA; Ratio (NGT/oral) = 0.987, 90% CI 2-sided [0.936 to 1.041]
Statistical Analysis 2: Comparison: MT-1186 Orally vs MT-1186 Via NGT; For AUC0-inf, MT-1186 orally Versus MT-1186 via NGT; Test type: Other — AUC0-inf was log-transformed and analyzed by analysis of variance using administration groups, the administration route, study periods, and subjects as factors. Estimates of the mean values on the log scale, the mean difference between administration routes on the log scale, and 90% CIs for the difference were back transformed to present mean ratios and their 90% CIs for administration via NGT to oral administration; ANOVA; Ratio (NGT/oral) = 0.981, 90% CI 2-sided [0.931 to 1.033]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Edaravone
Time Frame: Plasma samples are collected: Day 1 and Day 4 at pre-dose, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, and 12 hours; Day 2 and Day 5 at 24 and 36 hours; Day 3 and Day 6 at 48 hour after administration.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MT-1186 Orally | MT-1186 Via NGT
Number analyzed (Participants) | 36 | 36
ng/mL | 2470 (839.8) | 2775 (1444)
Statistical Analysis 1: Comparison: MT-1186 Orally vs MT-1186 Via NGT; MT-1186 orally Versus MT-1186 via NGT; Test type: Other — Cmax was log-transformed and analyzed by analysis of variance using administration groups, the administration route, study periods, and subjects as factors. Estimates of the mean values on the log scale, the mean difference between administration routes on the log scale, and 90% CIs for the difference were back transformed to present mean ratios and their 90% CIs for administration via NGT to oral administration; ANOVA; Ratio (NGT/oral) = 1.052, 90% CI 2-sided [0.903 to 1.227]

3. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Edaravone
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | MT-1186 Orally | MT-1186 Via NGT
Number analyzed (Participants) | 36 | 36
h | 0.50 [0.25 to 0.50] | 0.25 [0.08 to 1.00]

4. Primary Outcome: Terminal Elimination Half-life (t1/2) of Edaravone
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | MT-1186 Orally | MT-1186 Via NGT
Number analyzed (Participants) | 36 | 36
h | 21.52 (33.83) | 13.53 (13.81)

5. Primary Outcome: Apparent Terminal Elimination Rate Constant (Kel) of Edaravone
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | MT-1186 Orally | MT-1186 Via NGT
Number analyzed (Participants) | 36 | 36
1/h | 0.06430 (0.03776) | 0.07713 (0.03269)

6. Primary Outcome: Mean Residence Time (MRT) of Edaravone
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | MT-1186 Orally | MT-1186 Via NGT
Number analyzed (Participants) | 36 | 36
h | 4.66 (8.89) | 2.89 (1.44)

7. Primary Outcome: Apparent Total Clearance (CL/F) of Edaravone
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | MT-1186 Orally | MT-1186 Via NGT
Number analyzed (Participants) | 36 | 36
L/h | 42.8 (12.3) | 43.8 (12.6)

8. Primary Outcome: Apparent Distribution Volume at Elimination Phase (Vz/F) of Edaravone
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | MT-1186 Orally | MT-1186 Via NGT
Number analyzed (Participants) | 36 | 36
L | 1209 (1682) | 816 (782)

9. Primary Outcome: Apparent Distribution Volume at Steady State (Vss/F) of Edaravone
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | MT-1186 Orally | MT-1186 Via NGT
Number analyzed (Participants) | 36 | 36
L | 183.7 (299.9) | 125.4 (67.7)

10. Secondary Outcome: Number of Participants With Adverse Events and Adverse Drug Reactions
Time Frame: Day 1 to 11
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MT-1186 Orally | MT-1186 Via NGT
Number analyzed (Participants) | 36 | 36
Participants
  Number of Participants with Adverse events | 1 | 3
  Number of Participants with adverse drug reactions | 0 | 1

ADVERSE EVENTS:
Time Frame: The provision of informed consent to Day 11
Description: This study was designed as a 2-group, 2-period crossover study with the advance administration of edaravone orally group (Oral => NGT) with 18 subjects, and the advance administration of edaravone via NGT group (NGT => Oral) with 18 subjects to investigate the bioavailability between edaravone orally and via NGT.
Groups:
- MT-1186 Orally: Healthy subjects were administered a single dose of Edaravone oral suspension (105 mg) orally under fasted condition.
- MT-1186 Via NGT: Healthy subjects were administered a single dose of Edaravone oral suspension (105 mg) via NGT under fasted condition.
Arm/Group | MT-1186 Orally | MT-1186 Via NGT
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 1/36 | 3/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-1186 Orally (N=36) | MT-1186 Via NGT (N=36)
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT04776135/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT04776135/SAP_001.pdf